CLINICAL TRIAL: NCT02534805
Title: Patient Buddy App for the Prevention of Avoidable Readmission in Cirrhosis
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: HM20003950
Record Dates: First submitted 2015-08-05; First posted 2015-08-28 (Estimated); Results first posted 2025-07-17 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient Buddy: Subjects and caregivers will be given iphones loaded with the App that will be used to enter medications, issues and orientation questions. They will be seen at day 15 and day 30 and will receive a phone call day 7 and day 21 inquiring about issues that would need medical attention

SUMMARY:
To use the PatientBuddy App to reduce 30-day avoidable readmissions in cirrhotic patients using a patient and caregiver perspective.

DETAILED DESCRIPTION:
Specific aim 1: To perform a pilot and feasibility study of disseminating current knowledge of readmission prevention in cirrhosis by using the Patient Buddy App with patient and caregiver interfaces. Eighty subjects (40 cirrhotic inpatients and 40 caregivers) will be enrolled and trained on the Patient Buddy at discharge. The App focuses on daily communication between patient/caregivers and the study team based on previously identified risk factors associated with readmission. The study team will initiate measures to prevent readmission using these communications. A detailed analysis of 30-day readmissions and input of the patients,caregivers and nurse manager will be performed to improve the App. Avoidable readmissions will be defined by a committee of hepatologists who is not part of the study at VCU.

Specific aim 2: To incorporate the opinion of key stakeholders (patients, caregivers and case managers) towards improving the Patient Buddy App in the prevention of avoidable readmission in cirrhosis. The input of the key stakeholders and the analysis of readmissions prevented during the pilot study will be used to update the App for preventing avoidable readmissions in future studies

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis patients ≥21 years of age hospitalized for non-elective reasons
* Adult caregiver and the patient living in the same house
* Both (caregiver and patient) should be able to complete the Patient Buddy training and evaluation
* Discharged home from the hospital
* Patients who have VCU as a primary hospital base

Exclusion Criteria:

* Elective hospitalization
* Lack of an adult caregiver
* Active alcohol/substance abuse within 1 month of the hospitalization
* Unable to perform training or give consent
* Patients discharged to hospice, nursing home or extended care facilities
* Patients on Hemodialysis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic subjects who are hospitalized for non-elective reasons
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, Principal Investigator — VCU Medical Center
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Buddy Subject Only/Not Dyad: No dyads enrolled in this part of the study. Only the patients (subjects) were enrolled in this part of the study, not dyads. The numbers only represent the patient enrollment numbers. Patients were given iphones loaded with the Buddy App that was used to enter medications, issues and orientation questions. They were seen at day 15 and day 30 and received a phone call day 7 and day 21 inquiring about issues that would need medical attention.
- Standard of Care Subject Only/Not Dyad: No dyads enrolled in this part of the study. Subjects randomized to standard of care and not the Buddy App. Dyad unit not reported, only the patient/subject.
Period: Overall Study
Arm/Group | Patient Buddy Subject Only/Not Dyad | Standard of Care Subject Only/Not Dyad
Started | 116 | 116
Completed | 116 | 116
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only the patients (subjects) were enrolled in this part of the study, not dyads. The numbers only represent the patient subject enrollment numbers. Subjects were given phones loaded with the Buddy App, which was used to enter medications, issues, and orientation questions. They were seen on days 15 and 30 and received phone calls on days 7 and 21 inquiring about issues that would need medical attention.
Groups:
- Patient Buddy Subject Only/Not Dyad: Subjects will be given iphones loaded with the App that will be used to enter medications, issues and orientation questions. They will be seen at day 15 and day 30 and will receive a phone call day 7 and day 21 inquiring about issues that would need medical attention
- Standard of Care Subject Only/Not Dyad: Subjects randomized to standard of care and not the Buddy App
- Total: Total of all reporting groups
Arm/Group | Patient Buddy Subject Only/Not Dyad | Standard of Care Subject Only/Not Dyad | Total
Number analyzed (Participants) | 116 | 116 | 232
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (12.38) | 58.42 (8.89) | 58.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 40 | 98
  Male | 58 | 76 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 110 | 110 | 220
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 36 | 89
  White | 63 | 80 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 116 | 116 | 232

OUTCOME MEASURES:

1. Primary Outcome: Avoidable Readmission
Description: Avoidable Readmissions within 30 days.
Time Frame: 30 days
Measure: Number; unit: Number of Avoidable Readmissions
Groups:
- Patient Buddy Subject Only/Not Dyad: Only the patients (subjects) were enrolled in this part of the study, not dyads. The numbers only represent the subject enrollment numbers. Subjects were given phones loaded with the Buddy App, which was used to enter medications, issues, and orientation questions. They were seen on days 15 and 30 and received phone calls on days 7 and 21 inquiring about issues that would need medical attention.
- Standard of Care Subject Only/Not Dyad: Subjects randomized to standard of care and not the Buddy App. Just the patients counted and reported, not the dyads.
Arm/Group | Patient Buddy Subject Only/Not Dyad | Standard of Care Subject Only/Not Dyad
Number analyzed (Participants) | 116 | 116
Number of Avoidable Readmissions | 23 | 12

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Patient Buddy Subject Only/Not Dyad: Only the patients (subjects) were enrolled in this part of the study, not dyads. The numbers only represent the patient enrollment numbers. Patients were given phones loaded with the Buddy App, which was used to enter medications, issues, and orientation questions. They were seen on days 15 and 30 and received phone calls on days 7 and 21 inquiring about issues that would need medical attention.
Arm/Group | Patient Buddy Subject Only/Not Dyad | Standard of Care Subject Only/Not Dyad
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/116
Other Adverse Events (participants affected / at risk) | 0/116 | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT02534805/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT02534805/ICF_001.pdf